CLINICAL TRIAL: NCT01815853
Title: A Randomized, Open-Label, Multicenter, Controlled Phase III Trial Comparing Neoadjuvant Chemoradiotherapy Followed by Surgery and Adjuvant Chemotherapy Versus Neoadjuvant Chemotherapy Followed by Surgery and Adjuvant Chemotherapy in Patients With Locally Advanced Gastric Cancer
Brief Title: Neoadjuvant Chemoradiotherapy vs. Chemotherapy Followed by Radical Gastrectomy and Adjuvant Chemotherapy for Advanced Gastric Cancer
Acronym: Neo-CRAG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); Liaoning Cancer Hospital & Institute (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Zhejiang Cancer Hospital (Other); First Hospital of China Medical University (Other); The Affiliated Tumor Hospital of Guangxi Medical University (Unknown); Hangzhou First People's Hospital, School of Medicine, Zhejiang Universiry (Unknown); The Affiliated Hospital of Qingdao University (Other); Guangdong Provincial People's Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); National Clinical Research Center for Cancer/Cancer Hospital (Unknown)
Responsible Party: Principal Investigator, Zhou Zhiwei, Director of Gastric Surgery, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCCGPS2
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer
Keywords: Neoadjuvant; Chemoradiotherapy; Chemotherapy; Locally advanced gastric cancer; Pathological complete response; D2 gastrectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: Neoadjuvant Chemoradiotherapy versus Neoadjuvant Chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant Chemoradiotherapy (Experimental): Radiotherapy (45Gy/25f) + 3 cycles of XELOX Chemotherapy [Oxaliplatin 130 mg/m² IV on Day 1 + Capecitabine 1000 mg/m² orally BID on Days 1-14 of a 21-day cycle (non-concurrent); Oxaliplatin 100 mg/m² IV on Day 1 + Capecitabine 825 mg/m² orally BID on Days 1-14 of a 21-day cycle (concurrent chemoradiotherapy) ] following with D2 Gastrectomy and 3 cycles of Adjuvant XELOX Chemotherapy
  Interventions: Radiation: Neoadjuvant Chemoradiotherapy; Procedure: R0 D2 Gastrectomy; Drug: Adjuvant Chemotherapy
- Neoadjuvant Chemotherapy (Active Comparator): 3 cycles of XELOX Chemotherapy (Oxaliplatin 130 mg/m² IV on Day 1 + Capecitabine 1000 mg/m² orally BID on Days 1-14 of a 21-day cycle) following with D2 Gastrectomy and 3 cycles of Adjuvant XELOX Chemotherapy
  Interventions: Drug: Neoadjuvant Chemotherapy; Procedure: R0 D2 Gastrectomy; Drug: Adjuvant Chemotherapy

INTERVENTIONS:
Radiation: Neoadjuvant Chemoradiotherapy — Radiotherapy (45Gy/25f) + 3 cycles of XELOX Chemotherapy [Oxaliplatin 130 mg/m² IV on Day 1 + Capecitabine 1000 mg/m² orally BID on Days 1-14 of a 21-day cycle (non-concurrent); Oxaliplatin 100 mg/m² IV on Day 1 + Capecitabine 825 mg/m² orally BID on Days 1-14 of a 21-day cycle (concurrent chemoradiotherapy)]
  Arms: Neoadjuvant Chemoradiotherapy
Drug: Neoadjuvant Chemotherapy — 3 cycles of XELOX Chemotherapy (Oxaliplatin 130 mg/m² IV on Day 1 + Capecitabine 1000 mg/m² orally BID on Days 1-14 of a 21-day cycle)
  Arms: Neoadjuvant Chemotherapy
Procedure: R0 D2 Gastrectomy
Drug: Adjuvant Chemotherapy — 3 cycles of XELOX Chemotherapy (Oxaliplatin 130 mg/m² IV on Day 1 + Capecitabine 1000 mg/m² orally BID on Days 1-14 of a 21-day cycle)

SUMMARY:
Patients with histologically confirmed gastric adenocarcinoma with locally advanced gastric cancer are randomized in a 1:1 ratio to receive neoadjuvant chemoradiotherapy with DT45Gy/25f plus three cycles of XELOX therapy or neoadjuvant chemotherapy alone using XELOX regimen following D2 gastrectomy and adjuvant chemotherapy for 3 cycles. The primary end point is 3-year disease free survival (DFS), and secondary end point is 5-year overall survival (OS), R0 resection rate, pathological complete remission (pCR) and treatment safety.

DETAILED DESCRIPTION:
Background: Literatures have shown that patients with locally advanced gastric cancer could potentially benefit from neoadjuvant chemoradiotherapy, but whether this can improve patients' outcome is still unclear.

Patients and methods: In this study , patients with histologically confirmed gastric adenocarcinoma with pre-operative staging are cT3N2/N3M0, cT4aN+M0 and cT4bNanyM0, aged between 18-75 years old, with adequate organ function and having an Eastern Cooperative Oncology Group performance status score ≤2, are randomized in a 1:1 ratio to receive neoadjuvant chemoradiotherapy with DT45Gy/25f plus three cycles of XELOX therapy [Oxaliplatin 130 mg/m² IV on Day 1 + Capecitabine 1000 mg/m² orally BID on Days 1-14 of a 21-day cycle (non-concurrent); Oxaliplatin 100 mg/m² IV on Day 1 + Capecitabine 825 mg/m² orally BID on Days 1-14 of a 21-day cycle (concurrent chemoradiotherapy)] or neoadjuvant chemotherapy alone using XELOX regimen (Oxaliplatin 130 mg/m² IV on Day 1 + Capecitabine 1000 mg/m² orally BID on Days 1-14 of a 21-day cycle) following by D2 gastrectomy and adjuvant chemotherapy with same dosage of XELOX therapy for up to 3 cycles. The primary end point is 3-year disease free survival (DFS), and secondary end point is 5-year overall survival (OS), R0 resection rate, pathological complete remission (pCR) and treatment safety. The final study analytics are to be conducted at the end of the 5th year after the last patient's enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed gastric cancer with clinical staging determined by endoscopic ultrasound and contrast-enhanced CT or MRI as cT3N2/N3M0, cT4aN+M0, or cT4bNanyM0.
2. Good general condition, with Eastern Cooperative Oncology Group (ECOG) performance status <2 and no contraindications to surgery.
3. Ambulatory male or female patients aged 18 to 75 years.
4. Sufficient physical fitness and organ function to tolerate major abdominal surgery.
5. Baseline laboratory parameters meeting the following criteria: WBC > 4.0 × 10⁹/L, ANC > 1.5 × 10⁹/L, Hb ≥ 100 g/L, PLT ≥ 100 × 10⁹/L, total bilirubin ≤ 1.5 × upper limit of normal (ULN), AST and ALT ≤ 2.5 × ULN, and serum creatinine ≤ 1.0 × ULN.
6. No prior or concurrent diagnosis of other malignancies.
7. Willing and able to comply with study protocol requirements during the trial period.
8. Provided written informed consent prior to screening, with full awareness of the right to withdraw from the study at any time without consequence.
9. Estimated life expectancy of at least 3 months.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or women of childbearing potential not using effective contraception.
2. Receipt of any antitumor therapy prior to surgery.
3. History of or concurrent malignancies other than gastric cancer.
4. Presence of psychiatric disorders, brain metastases, or leptomeningeal metastases.
5. Uncontrolled or severe comorbid conditions or active infections.
6. Decompensated dysfunction of major organs (e.g., cardiac, pulmonary, hepatic, or renal failure).
7. Concurrent participation in another clinical trial.
8. Contraindications to chemotherapy, radiotherapy, or surgery.
9. Active hepatitis B or hepatitis C virus infection.
10. Grade ≥2 peripheral neuropathy (per NCI-CTCAE).
11. Chronic intestinal diseases or short bowel syndrome.
12. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
13. Known hypersensitivity to capecitabine or any of its excipients.
14. Ongoing treatment with sorivudine or related analogs.
15. Deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2025-06 (Actual); Study Completion 2025-06 (Actual)

PRIMARY OUTCOMES:
Disease-free Survival | 3 years
  3-year DFS

SECONDARY OUTCOMES:
Overall Survival | 5 years
  5-year Overall Survival
Pathological Complete Remission | Peri-operative period
  pCR
Radical Resection Rate | Peri-operative period
  R0 Resection Rate
Adverse effects | Peri-operative period
  Treatment safety

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-wei Zhou, M.D, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China